CLINICAL TRIAL: NCT00126451
Title: A Phase II Clinical Study of Oral Suberoylanilide Hydroxamic Acid in Patients With Relapsed or Refractory Breast, Colorectal, and Non-small Cell Lung Cancer.
Brief Title: A Clinical Trial of Oral Suberoylanilide Hydroxamic Acid (SAHA) in Patients With Relapsed or Refractory Breast, Colorectal and Non-Small Cell Lung Cancer (0683-011)(TERMINATED)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0683-011; 2005_014
Record Dates: First submitted 2005-08-02; First posted 2005-08-04 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Breast Cancer; Colorectal Cancer; Non-small-cell Lung Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Vorinostat; RE1-silencing transcription factor

INTERVENTIONS:
Drug: MK0683, vorinostat, Suberoylanilide Hydroxamic Acid (SAHA)
Drug: Duration of Treatment - During each treatment cycle, treatment is administered twice daily for 14 days, followed by 7 days of rest for a total of 10 cycles

SUMMARY:
This is an investigational study to determine the response rate of relapsed/refractory breast, colorectal and non-small cell lung cancer to oral suberoylanilide hydroxamic acid (SAHA), to evaluate PET as an earlier indicator of response to SAHA as assessed by response evaluation criteria in solid tumours (RECIST) criteria and to evaluate the safety and tolerability of oral suberoylanilide hydroxamic acid.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 18 years or older with confirmed diagnosis of breast adenocarcinoma, colorectal carcinoma or non-small cell lung cancer
* Patients must have relapsed or refractory disease following at least one chemotherapeutic treatment regimen.
* Has a measurable, positron emission tomography (PET) assessable lesion
* Adequate blood, liver, bone marrow and kidney functions
* Has not received any chemotherapy for at least 4 weeks prior to entry in this study
* Agrees to take adequate measures to prevent pregnancy.

Exclusion Criteria:

* Patient has had prior treatment with histone deacetylase (HDAC) inhibitor.
* Patient has had treatment with investigational agents within the last 30 days.
* Patient has active infection or had intravenous (IV) antibiotic, antiviral, or antifungal medications within 2 weeks of the start of study drugs.
* Patient has HIV, hepatitis B or hepatitis C infection.
* Patient is pregnant or lactating.
* Patient has allergy to any component of the study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2004-12-01 (Actual); Primary Completion 2005-10-11 (Actual); Study Completion 2005-10-11 (Actual)

PRIMARY OUTCOMES:
Response rate of relapsed/refractory breast, colorectal and non-small cell lung cancer to SAHA using RECIST criteria.

SECONDARY OUTCOMES:
Positron emission tomography (PET) as an earlier indicator of the response to SAHA as assessed by RECIST criteria. To evaluate the safety and tolerability of SAHA for 14 days every 21 days.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Vansteenkiste J, Van Cutsem E, Dumez H, Chen C, Ricker JL, Randolph SS, Schoffski P. Early phase II trial of oral vorinostat in relapsed or refractory breast, colorectal, or non-small cell lung cancer. Invest New Drugs. 2008 Oct;26(5):483-8. doi: 10.1007/s10637-008-9131-6. Epub 2008 Apr 19. PMID 18425418
- Available data/document: CSR Synopsis Link — http://www.merck.com/clinical-trials/policies-perspectives.html